CLINICAL TRIAL: NCT00698984
Title: Pilot Study To Investigate The Effect Of Bonistein(R) Bone Blend Containing Genistein, Polyunsaturated Fatty Acids (N-3 PUFAS) And Vitamins K1 And D3 On Bone Mineral Density (BMD), Bone Mineral Content (BMC) And Biomarkers Of Bone Health In Early Postmenopausal Women
Brief Title: Investigation of the Effect of BONISTEIN(R) Bone Blend on Bone Mineral Density/Content and Biomarkers of Bone Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Robert P. Heaney, Creighton University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GEN/BLEND-06.06
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2009-01-16 (Estimated); Status verified 2009-01

CONDITIONS: Osteoporosis
Keywords: Soy Isoflavones, Bone Mineral Density, Bone Mineral Content, postmenopausal Women, Bone Markers, Bone Health, Phytoestrogens
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 30 mg BONISTEIN(R) 150 ug Vitamin K1 800 IU Vitamin D3 1000 mg PUFA 500 mg Calcium
  Interventions: Dietary Supplement: BONISTEIN(R) bone blend
- 2 (Placebo Comparator): 500 mg Calcium
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: BONISTEIN(R) bone blend — 2 Capsules per day over a period of 6 months
  Arms: 1
Dietary Supplement: Placebo — 2 capsules per day over a period of 6 months
  Arms: 2

SUMMARY:
The purpose of this study is to obtain information about the effect of a combination of genistein, PUFAs, vitamin K and D (BONISTEIN(R) bone blend) on bone health, determined as bone mass density/content and bone biomarkers after 6-months treatment in 70 healthy postmenopausal women. In addition, safety and tolerability will be investigated.

DETAILED DESCRIPTION:
Osteoporosis is the most frequent disease of the skeletal system with approximately one third of all postmenopausal women being currently affected in the USA and in Europe. The role of nutrition in bone health has been increasingly recognized in the last couple of years. In particular nutrients such as isoflavones, vitamins D and K as well as polyunsaturated fatty acids (PUFA) have been implicate in bone health recently.

The DSM Nutritional Products Ltd product BONISTEIN(R) is a synthetic genistein. Its genistin aglycone purity is above 99 % and the appearance is a beige crystal.

In addition to the primary and secondary outcomes, body composition, genistein plasma levels, diet and physical activity are assessed.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 45 (inclusive) to 55 years (inclusive)
* Race: Caucasian
* Non-smokers / Smokers up to 10 cigarettes/day
* Postmenopausal hormone status: 1-3 years since the last spontaneous menstrual bleeding and a follicle-stimulating hormone concentration (FSH) >75 IU/ml and 17-estradiol (E2) of < 20 ng/L
* Years since menopause between 1-3 years
* Natural menopause or total hysterectomy with bilateral salpingo-oophorectomy
* Subjects with E2 results within the inclusion criteria range will be assessed on an individual basis if FSH level is less than 75 IU/ml
* Assessed as age-related healthy, based on a pre-study examination including medical history, physical examination, ECG, vital signs and clinical laboratory. The examination will be performed by a MD at the study site within 1-2 months prior planned study start for the individual subject.
* Willingness and ability to give written informed consent and willingness and ability to understand, to participate and to comply with the study requirements.
* Ability to understand, speak, read and write the English language

Exclusion Criteria:

* T-score < -2.5 at total hip and spine (either or both)
* Suspect lack of compliance
* BMI > 30 or < 21
* Use of HRT within the previous 6 months
* Use of any drug which might interfere with bone-metabolism (bisphosphate, estrogen receptor modulators, calcitonin) within the previous 12 months
* Systematic practice of high intensity exercise
* Vegetarian nutrition or any other extreme dietary habits
* Use of dietary supplements while on study, except multi vitamin. No "wash out" period for supplements - must stop before run-in period and refrain until the end of the study.
* Participant in any other study or donation of blood during the last 30 days before start of each dosing phase (T0).
* Total genistein blood concentrations of > 100 ng/ml measured at pre-study examination
* Known hypersensitivity or allergy to soy, purified isoflavones, peanuts, fish, and/or genistein.
* Hepatitis screen (serology) positive or not performed
* Drug screen positive or not performed (at least amphetamines, benzodiazepines, cannabinoides, opiates).
* Subjects on a weight reduction program or a medically supervised diet
* Unexplained weight loss or weight gain of more than 5 kg in the three months prior to the study
* History of liver or pancreas diseases
* Cardiovascular diseases, even AV-block I0 (PQ time > 220 ms) and QTc time > 450 ms
* History of breast cancer, endometrial cancer and other malignancy except basal and squamous cell skin cancer
* History of thromboembolism or deep venous thrombosis
* Any fractures within one year except for fingers, toes and facial bones
* Subjects with susceptibility for fractures as a history of being a faller
* Endometrial thickness > 6 mm
* Endometrial polyps
* Untreated hypo- or hyperthyroidism
* Insulin-dependent diabetes mellitus, Crohn's Disease, Cushing Disease etc.
* Any condition which might interfere with absorption of the investigational product (e.g. malabsorption syndrome)
* Co-medication: Anticoagulants, parathyroid hormones, corticosteroids, thiazide diuretic
* Subjects who, during the previous 24 months, received a total fee payment greater than 5'000 USD for participation in biomedical research

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density/Content (BMD/BMC) at lumbar spine and femoral neck | Baseline and after 6 months

SECONDARY OUTCOMES:
BMD/BMC on whole body, Ward's Triangle, total hip, and (inter)trochanter Bone resorption markers: DPD, NTX, RANKL/OPG Bone formation markers: bALP, OC, ucOC | Baseline and after 3 and 6 months (bone markers)

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Heaney, MD, Principal Investigator — Creighton University Medical Center - Osteoporosis Research Center
Locations (1):
- Creighton University Medical Center - Osteoporosis Research Center, Omaha, Nebraska, United States